CLINICAL TRIAL: NCT02142439
Title: Strength Training and Eating Disorders (STERK - Styrketrening og Spiseforstyrrelser)
Brief Title: STERK - Strength Training and Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Collaborators: University of Agder (Other); Norwegian School of Sport Sciences (Other); Modum Bad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STERK
Record Dates: First submitted 2014-02-27; First posted 2014-05-20 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Eating Disorders
Keywords: Anorexia; Bulimia; Physical activity; Treatment
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia; Bulimia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention group 1 (Experimental): Exercise counseling 1 time/week, Strength training 3 times/week, dose: 5 RM x 3 sets.
  Interventions: Behavioral: Strength training
- Intervention group 2 (Experimental): Exercise counseling 1 time/week. Strength training 3 times/week, dose: 10 RM x 3 sets.
  Interventions: Behavioral: Strength training
- Intervention group 3 (Experimental): Exercise counseling 1 time/week. Strength training 3 times/week, dose: 30 RM x 3 sets
  Interventions: Behavioral: Strength training
- Control group (No Intervention): Exercise counseling 1 time/week

INTERVENTIONS:
Behavioral: Strength training — Three times per week with strength training
  Arms: Intervention group 1; Intervention group 2; Intervention group 3

SUMMARY:
Strength training has been found effective for enhancement of bone health, muscle strength and body composition among premenopausal women from the general population, however it is unclear to what extend strength training might improve these parameters among women with eating disorders. The aim of this study is therefore to examine acute and long-term effects of strength training among persons with eating disorders. The study is a randomized, controlled, single-blinded trial with three intervention groups and one control group. The three intervention groups will perform different volumes of strength training. The intervention period is 16 weeks with three sessions per week. At pretest, posttest, and 6 months, 12 months and 24 months follow-up, the following variables will be measured: bone health, muscle strength, power, body composition hormone levels, physical activity level and compulsivity, body awareness, quality of life, and eating disorders psychopathology. Qualitative in-depth interviews will be carried out to explore the participants' experiences with strength training. The study is carried out in Norway, and is performed in collaboration with Telemark University College, University of Agder, Norwegian school of sport sciences and Modum Bad psychiatric center. The results from the study might implicate on strength training as part of treatment for eating disorders.

DETAILED DESCRIPTION:
ED are mental disorders which often lead to serious medical complications such as hormone disturbances, osteopenia/osteoporosis, and myopathy. More than 90% of females with anorexia nervosa (AN) have osteopenia, and almost 40% have osteoporosis. Osteoporosis in the European Union is estimated to cost 37 billion euros each year, and the majority of persons with osteoporosis are untreated. Although economic analysis of osteoporosis in Norway is lacking, the prevalence of osteoporosis in Norway is among the world's highest.

Strength training is effective in treatment of osteoporosis among postmenopausal women. Despite this, evidence based knowledge about strength training as a possible treatment-option for osteopenia/osteoporosis in ED is lacking. Due to the long half-life of bisphosphonates, such medications must be used carefully among young adults. Hence, there are no current well-documented treatment strategies for osteopenia/osteoporosis for this age group.

Although excessive physical activity is a common symptom among persons with ED, strength training is an exercise modality rarely used in this population. In addition, restoration of body weight is an important treatment goal for underweight persons with ED. Such a weight restoration leads to altered body composition with higher increase in adipose tissue compared to lean tissue, and the adipose tissue often redistribute to more abdominal fat. Such altered body composition might increase risk of cardiovascular disease and increased body dissatisfaction, and hence increase risk of relapse.

Strength training affects body composition in persons both with and without ED. It is therefore interesting to examine if strength training intervention affects body dissatisfaction, and hence reduce psychopathology and increase quality of life, among persons suffering from ED.

Existing studies with strength training intervention use different repetitions, sets and intensities. Campos et al. found that few repetitions (i.e. 3-5 rep x 3 sets) were more effective in increasing muscle strength compared to medium (9-11 rep x 3) and many repetitions (20-28 rep x 2), while the latter gave largest increase in muscular endurance among healthy males. Mosti et al. found increased bone mass in lumbar spine and femur neck and alterations in blood bone markers after 12 weeks of strength training (3-5 reps x 4 sets, 85-90% of 1RM) among postmenopausal women with osteopenia/osteoporosis. A study using both low and high intensity strength training intervention lasting for 12 months found increased bone mineral density (BMD) in lumbar spine among healthy elderly women. The few existing studies using strength training among persons with ED have all used low intensity strength training, and none of these have examined the effects on bone health. Two randomized controlled trials found effect of strength training on body composition, muscle strength and quality of life among persons with Anorexia Nervosa, whereas Del Valle et al. only found effects on quality of life. The low intensity might explain the lack of effects in the latter study. It is therefore a need for studies using adequate dosage of strength training among persons with ED.

Strength training is a treatment method with few possible side effects. Such training might however lead to a drop in blood pressure, this is a possible side effect among persons with ED because hypotension is more prevalent in this population compared to the general population. Due to safety reasons, this aspect is important to map.

Approaches, hypotheses and choice of method

The following research questions problems (RQ) have been defined:

RQ 1: What is the effect of different strength training regimes on bone health among persons with ED? RQ 2: What is the effect of different strength training regimes on body composition, hormone levels, muscle strength and power among persons with ED? RQ 3: What is the effect of different strength training regimes on ED psychopathology, body awareness and quality of life among persons with ED? RQ 4: What is the effect of different strength training regimes on weekly physical activity, motives for physical activity and compulsive exercise among persons with ED? RQ 5: What is the immediate effect of different strength training regimes on blood pressure among persons with ED? RQ 6: How do persons with ED experience the use of strength training as part of treatment for ED? RQ 7: What is the long-term effect of different strength training regimes on bone health among persons with ED? RQ 8: What is the long-term effect of different strength training regimes on body composition, hormone levels, muscle strength and power among persons with ED? RQ 9: What is the long-term effect of different strength training regimes on ED psychopathology, body awareness and quality of life among persons with ED? RQ 10: What is the long-term effect of different strength training regimes on weekly physical activity, motives for physical activity and compulsive exercise among persons with ED?

To examine the research questions, we will use a multi-methods approach. We will conduct a randomized controlled trial with four groups (n=200), these groups will be followed during the 16 weeks intervention period and up to two years follow-up. We will use both quantitative objective and self-report assessment methods, and qualitative in-depth interviews. To answer RQ 1 and RQ 2, objective assessment methods such as dual x-ray absorptiometry (DXA), blood samples and strength tests using squats and bench press will be conducted. RQ 3 and RQ 4 are answered by using standardized self-report instruments. Ambulatory continuous blood pressure monitors will be used during the first strength training session to answer RQ 5. RQ 6 will be answered by selecting participants to be informants in a qualitative semi-structured in-depth interview. To answer RQ 7-10, follow-up 6 months, 12 months and 24 months after the intervention will be conducted. We have chosen a randomized controlled design because it is the gold standard when examining effects of different treatment interventions. However, we believe it is important to take the participants' experiences into account, because this can give valuable additional information about the clinical significance of the interventions. Such information is valuable when considering the use of strength training intervention in clinical settings in the future. In evidence-based practice, it is essential to considerate both clinical expertise, a wide research perspective and the patients' preferences and subjective experiences of needs. This justify the use of a multi-methods approach where both quantitative objective and qualitative data are included.

Bone health is promoted through regular weight-bearing physical activity that use muscular strength and power and exert force on the skeleton above normal amounts. This project will expand the knowledge about how strength training can be used as a component of treatment in ED. Strength training has several benefits for persons with and without ED, however the existing studies have not examined one of the most important parameters, i.e. bone health. This project therefore seeks to assess parameters which allow us to explore the effects of strength training in details. Furthermore, we will examine and take the participants' own experiences into account. This is important so that future treatment can design and adapt the exercises to each individual.

ELIGIBILITY:
Inclusion Criteria:

* Meeting diagnostic criteria for anorexia nervosa, bulimia nervosa or eating disorders not otherwise specified
* Outpatient/home-dwelling
* Age: 18 years or older
* Premenopausal women

Exclusion Criteria:

* BMI <15 kg/m2
* Osteoporosis (t-score < -2,5 including low energy fracture)
* Psychosis, suicidal behavior
* Planned changes in medication during the 16 weeks of intervention
* Planned pregnancy within the 16 weeks intervention period, and/or up to one year follow-up (due to DXA scanning)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (DXA) | up to two years follow-up

SECONDARY OUTCOMES:
1RM squats | 16 weeks, two years follow-up
  1 repetition maximum (RM) for lower extremities (squats) and upper extremities (bench press)
1RM bench press | 16 weeks, two years follow-up
  1 repetition maximum (RM) for lower extremities (squats) and upper extremities (bench press)
Eating Disorders Examination clinical interview | 16 weeks, two years follow-up
  Clinical interview using Eating Disorders Examination Interview
DXA | 16 weeks, two years follow-up
  Measure body weight, and lean body mass and adipose tissue by DXA
Self-reported physical activity behavior | 16 weeks, two years follow-up
  Assess physical activity volume (duration, frequency and intensity) through exercise log Assess compulsivity through Compulsive Exercise Test
symptom check list (SCL-90) | 16 weeks, two years follow-up
  General psychopathology
Hormone levels | 16 weeks, two years follow-up
  Blood sample of Insuline Growth Factor (IGF-1), Thyroid stimulating hormone (TSH), T3, T4, leptine, cortisol, estradiol, progesterone, growth hormone (GH)
blood levels | 16 weeks, two years follow-up
  Calcium, vit D, sodium, potassium, magnesium, phosphate, blood sugar and cholesterol

OTHER OUTCOMES:
Body attitude | 16 weeks, two years follow-up
  Body Attitudes Test
Short Form - 36 | 16 weeks, two years follow-up
  Quality of life
Participants' experience with strength training | 16 weeks
  In-depth qualitative interview

CONTACTS AND LOCATIONS:
Overall Officials: Solfrid Bratland-Sanda, PhD, Study Chair — University of South-Eastern Norway
Locations (3):
- Norway (3):
  - University of Agder, Kristiansand, Agder
  - Telemark University College, Bø, Telemark
  - Norwegian school of sport sciences, Oslo

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available to other researchers

REFERENCES:
- [Background] Shroff H, Reba L, Thornton LM, Tozzi F, Klump KL, Berrettini WH, Brandt H, Crawford S, Crow S, Fichter MM, Goldman D, Halmi KA, Johnson C, Kaplan AS, Keel P, LaVia M, Mitchell J, Rotondo A, Strober M, Treasure J, Woodside DB, Kaye WH, Bulik CM. Features associated with excessive exercise in women with eating disorders. Int J Eat Disord. 2006 Sep;39(6):454-61. doi: 10.1002/eat.20247. PMID 16637047
- [Background] Mehler PS, Cleary BS, Gaudiani JL. Osteoporosis in anorexia nervosa. Eat Disord. 2011 Mar-Apr;19(2):194-202. doi: 10.1080/10640266.2011.551636. PMID 21360368
- [Background] Grinspoon S, Thomas E, Pitts S, Gross E, Mickley D, Miller K, Herzog D, Klibanski A. Prevalence and predictive factors for regional osteopenia in women with anorexia nervosa. Ann Intern Med. 2000 Nov 21;133(10):790-4. doi: 10.7326/0003-4819-133-10-200011210-00011. PMID 11085841
- [Background] Borer KT. Physical activity in the prevention and amelioration of osteoporosis in women : interaction of mechanical, hormonal and dietary factors. Sports Med. 2005;35(9):779-830. doi: 10.2165/00007256-200535090-00004. PMID 16138787
- [Background] Mosti MP, Kaehler N, Stunes AK, Hoff J, Syversen U. Maximal strength training in postmenopausal women with osteoporosis or osteopenia. J Strength Cond Res. 2013 Oct;27(10):2879-86. doi: 10.1519/JSC.0b013e318280d4e2. PMID 23287836
- [Background] Szabo CP, Green K. Hospitalized anorexics and resistance training: impact on body composition and psychological well-being. A preliminary study. Eat Weight Disord. 2002 Dec;7(4):293-7. doi: 10.1007/BF03324975. PMID 12588057
- [Background] Chantler I, Szabo CP, Green K. Muscular strength changes in hospitalized anorexic patients after an eight week resistance training program. Int J Sports Med. 2006 Aug;27(8):660-5. doi: 10.1055/s-2005-865812. PMID 16874594